CLINICAL TRIAL: NCT03619005
Title: Prasterone (DHEA) for the Treatment of Hypoactive Sexual Desire Disorder (HSDD) - Second Study (Placebo-Controlled, Double-Blind and Randomized Phase III Study of Intravaginal Prasterone)
Brief Title: Prasterone (DHEA) for the Treatment of Hypoactive Sexual Desire Disorder (HSDD) - Second Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision to not continue this study (only few subjects were screened).
Sponsor: EndoCeutics Inc. (Industry)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-245
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Hypoactive Sexual Desire Disorder (HSDD)
Keywords: Prasterone; DHEA; Menopause; Sexual Disorder; HSDD
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Vaginal Insert
- Prasterone (Active Comparator)
  Interventions: Drug: Prasterone 6.5 mg (0.50%) Vaginal Insert

INTERVENTIONS:
Drug: Placebo Vaginal Insert — Daily administration of a placebo vaginal insert.
  Arms: Placebo
Drug: Prasterone 6.5 mg (0.50%) Vaginal Insert — Daily administration of a 6.5 mg (0.50%) prasterone vaginal insert.
  Arms: Prasterone

SUMMARY:
The primary objective is to confirm the efficacy of intravaginal prasterone (DHEA) on Hypoactive Sexual Desire Disorder (HSDD) in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria (main criteria):

* Postmenopausal women (hysterectomized or not).
* Women between 40 and 80 years of age.
* Being in a stable relationship with the opportunity for sexual activity or masturbation at least once a month during the last 6 months or longer (before screening visit) and during the following 8 months.
* Diagnosis of HSDD confirmed by a qualified clinician.
* Willing to participate in the study and sign an informed consent.

Exclusion Criteria (main criteria):

* Chronic or acute life stress or major life change that could have interfered and continues to interfere significantly with sexual activity.
* Taking drugs which could be responsible for HSDD.
* Severe medical condition which can explain the loss of sexual desire.
* The administration of any investigational drug within 30 days of screening visit.
* Clinically significant abnormal serum biochemistry, urinalysis or hematology.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Sexual desire | 28 weeks
  Change from Baseline in sexual desire as evaluated by Questions 1 & 2 of the 19-items questionnaire titled Female Sexual Function Index (FSFI). For this outcome, Question 1 and Question 2 (corresponding to the desire domain) will be graded from 1 to 5 (score range) and then be multiplied by 0.6 (domain factor). The desire domain (sum of scores from Questions 1 & 2) has a minimum score of 1.2 and a maximum score of 6. Higher values represent a better outcome.
Distress from low sexual desire | 28 weeks
  Change from Baseline in distress from low sexual desire as evaluated by Question 13 of the 15-items questionnaire titled Female Sexual Distress Scale - Desire Arousal Orgasm (FSDS-DAO). For this outcome, Question 13 is graded from 0 to 4 and a lower value represents a better outcome.

SECONDARY OUTCOMES:
Satisfying sexual events (SSEs) | 28 weeks
  Change from Baseline in the number of SSEs from a daily log of sexual activity.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Labrie, M.D., Ph.D., Study Chair — EndoCeutics Inc.
Locations (10):
- United States (10):
  - Endoceutics site # 106, Huntsville, Alabama
  - Endoceutics site # 17, San Diego, California
  - Endoceutics site # 125, New London, Connecticut
  - Endoceutics site # 114, St. Petersburg, Florida
  - Endoceutics site # 119, Roswell, Georgia
  - Endoceutics site # 91, Savannah, Georgia
  - Endoceutics site # 20, New York, New York
  - Endoceutics site # 115, Fargo, North Dakota
  - Endoceutics site # 127, Bluffton, South Carolina
  - Endoceutics site # 102, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Labrie F, Archer D, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Berger L, Gilbert L, Martel C, Balser J. Effect of intravaginal dehydroepiandrosterone (Prasterone) on libido and sexual dysfunction in postmenopausal women. Menopause. 2009 Sep-Oct;16(5):923-31. doi: 10.1097/gme.0b013e31819e85c6. PMID 19424093
- [Background] Labrie F, Derogatis L, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; Members of the VVA Prasterone Research Group. Effect of Intravaginal Prasterone on Sexual Dysfunction in Postmenopausal Women with Vulvovaginal Atrophy. J Sex Med. 2015 Dec;12(12):2401-12. doi: 10.1111/jsm.13045. Epub 2015 Nov 23. PMID 26597311
- [Background] Bouchard C, Labrie F, Derogatis L, Girard G, Ayotte N, Gallagher J, Cusan L, Archer DF, Portman D, Lavoie L, Beauregard A, Cote I, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Group. Effect of intravaginal dehydroepiandrosterone (DHEA) on the female sexual function in postmenopausal women: ERC-230 open-label study. Horm Mol Biol Clin Investig. 2016 Mar;25(3):181-90. doi: 10.1515/hmbci-2015-0044. PMID 26725467